CLINICAL TRIAL: NCT04017078
Title: Assessment of Carotid Artery Calcifications on Digital Panoramic Radiographs and Its Relationship wıth Periodontal Condition and Cardiovascular Risk Factors
Brief Title: Assessment of Carotid Artery Calcifications
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, Assosc.Prof.Ph.D, Baskent University
Other Study IDs: MCetin
Record Dates: First submitted 2019-06-27; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Carotid Artery Calcification; Periodontal Diseases
Keywords: carotid artery calcification; panoramic radiography; periodontitis; periodontal disease; systemic diseases
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who referred for periodontal therapy: Patients who referred to Baskent University, Faculty of Dentistry, Department of Periodontology, during 2016-2018
  Interventions: Other: diagnosis of carotid artery calcification on digital panoramic radiograph

INTERVENTIONS:
Other: diagnosis of carotid artery calcification on digital panoramic radiograph — Suspected carotid arty calcifications findings were defined as one or more radiopaque mass adjacent to the cervical vertebrae at or below the intervertebral space between C3 and C4 on the DPR.

SUMMARY:
The aim of the study was to determine retrospectively the presence of carotid artery calcification (CAC) detected on digital panoramic radiographs (DPRs) and correlate the finding of such calcifications with gender, smoking status, medical history and periodontal status.The authors hypothesized that more CACs could observed in DPRs of individuals with periodontitis and CACs may correlate with the various risk factors included age, gender, smoking status, medical history.DPRs, periodontal status, medical (hypertension, diabetes, hyperlipidemia, cardiovascular disease) and smoking stories of 1101 patients (576 males, 525 females) were evaluated. The patients were divided into two groups as CAC detected in dental DPRs [CAC(+)] and those who were not [CAC (-)]. Periodontal status categorized as gingivitis, periodontitis and gingivitis with reduced periodontium.

DETAILED DESCRIPTION:
The first aim of the study was to determine retrospectively the presence of CACs detected on digital panoramic radiographs (DPRs) and second to correlate the finding of such calcifications with gender, smoking status, medical history and periodontal status. The authors hypothesized that more CACs could observed in DPRs of individuals with periodontitis and CACs may correlate with the various risk factors included age, gender, smoking status, medical history.

DPRs, periodontal status and medical stories of 1101 patients (576 males, 525 females) referred to Baskent University, Faculty of Dentistry, Department of Periodontology, during 2016-2018 were evaluated in this retrospective, cross-sectional study. This study was approved by Baskent University Institutional Review Board and supported by Baskent University Research Fund. All study procedures were performed in accordance with the Declaration of Helsinki and Research Committee Regulations.

Medical histories included gender, age, hypertension, diabetes, cardiovascular diseases, hyperlipidemia and smoking status. All data were obtained from the hospital records of the patients. Periodontal status of the participants also were determined based on hospital records.

All digital panoramic images were acquired using the same machine , with the following exposure parameters: 64-66 kVp; 6-9 mA; and 10 s. An observer with 7 years of experience at the Dentomaxillofacial Radiology department of the investigator's university evaluated the images on 2 different dates and 30 days apart by using the ClearCanvas program on an LED monitor under low light. Suspected CACs findings were defined as one or more radiopaque mass adjacent to the cervical vertebrae at or below the intervertebral space between C3 and C4 on the DPR .18 The CAC's were scored as present (+) or absent (-) by the dentomaxillofacial radiologist.Statistical analysis Whether the distributions of continuous variables were normally or not being determined by Kolmogorov Smirnov test. Levene test was used for the evaluation of homogeneity of variances. While, categorical data were shown as number of cases and percentages, otherwise, descriptive statistics for continuous variables were expressed as mean ± SD or median (min-max) percentiles, where applicable.

While, the mean differences between groups were compared by Student's t test, otherwise, Mann Whitney U test was applied for comparisons of not normally distributed data. Categorical data were analyzed by Continuity Corrected Chi-square or Fisher's Exact test, where appropriate.

Determining the best predictor(s) which effect on the existence of carotid artery calcification was evaluated by Multiple Logistic Regression Analysis. Any variable whose univariable test had a p value <0.25 was accepted as a candidate for the multivariable model along with all variables of known clinical importance. Odds ratios, 95% confidence intervals and Wald statistic for each independent variable were also calculated.Data analysis was performed by using IBM SPSS Statistics version 17.0 software. p value less than 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to Baskent University, Faculty of Dentistry, Department of Periodontology, during 2016-2018

Exclusion Criteria:

* Subjects with the lack of medical data
* DPRs not showing vertebra C3 and C4 were excluded.

Ages: 14 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Baskent University, Faculty of Dentistry, Department of Periodontology
Sampling Method: Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
prevalance of carotid artery calcifications | The images were evaluated in two months.
  Suspected CACs findings were defined as one or more radiopaque mass adjacent to the cervical vertebrae at or below the intervertebral space between C3 and C4 on the DPR.The CAC's were scored as present (+) or absent (-) by the dentomaxillofacial radiologist.

SECONDARY OUTCOMES:
The medical data of the patients with and without suspected CACs. | Medical data was recorded in two months.
  All medical data were obtained from the hospital records.if the patient was taking medication for hypertension, he was noted as a hypertensive patient. if the patient was taking medication for diabetes, he was noted as a patient with diabetes.If the patient was taking medication for hyperlipidemia, he was noted as a patient with hyperlipidemia.according to smoking status patients divided into three groups as never smoked, current smokers, former smokers.
Bleeding on probing (BOP)values of the patients with and without suspected CACs. | BOP values were recorded in two months.
  On periodontal examination, bleeding on probing (BOP) were evaluated in each patient. All periodontal measurements were recorded at six sites around each tooth by a periodontal probe excluding third molar.
Probing pocket depth (PPD) of the patients with and without suspected CACs. | PPD values were recorded in two months.
  Probing pocket depth (PPD = distance between gingival margin and bottom of the periodontal pocket)were evaluated in each patient. All periodontal measurements were recorded at six sites around each tooth by a periodontal probe excluding third molar.
Clinical attachment level (CAL of the patients with and without suspected CACs. | CAL values were recorded in two months.
  Clinical attachment level (CAL = distance between the cemento-enamel junction and bottom of the periodontal pocket)were evaluated in each patient. All periodontal measurements were recorded at six sites around each tooth by a periodontal probe excluding third molar.
Periodontal status of the patients with andwithout suspected CACs. | Periodontal status was recorded in two months.
  Periodontal status was categorized as gingivitis, reduced periodontium with gingivitis and periodontitis. When no clinical attachment loss and/or recession, probing depths 3 mm or less, BOP ≥ %10 of sites were present, the diagnosis was gingivitis. If gingival inflammation was noted with clinical attachment loss and/or recession, probing depths ≤ 3 mm, BOP ≥ %10 of sites, the patient was diagnosed as reduced periodontium with gingivitis. The patients who had interdental CAL at ≥ 2 non-adjacent teeth or buccal or oral CAL ≥ 3 mm with probing depths >3 mm at ≥ 2 teeth and BOP ≥ %10 of sites were diagnosed as periodontitis.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Bilgin Çetin, DDS,PhD, Principal Investigator — Department of Periodontology, Faculty of Dentistry, Baskent University
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilgin Cetin M, Sezgin Y, Nisanci Yilmaz MN, Koseoglu Secgin C. Assessment of carotid artery calcifications on digital panoramic radiographs and their relationship with periodontal condition and cardiovascular risk factors. Int Dent J. 2020 Sep 29;71(2):160-6. doi: 10.1111/idj.12618. Online ahead of print. PMID 32996164